CLINICAL TRIAL: NCT04363697
Title: A Multicenter, Randomized, Double-Blind, Parallel Group, Placebo-Controlled Trial to Evaluate the Effect of In-Hospital Initiation of Dapagliflozin on Clinical Outcomes in Patients Who Have Been Stabilized During Hospitalization for Acute Heart Failure DAPAgliflozin and Effect on Cardiovascular Events in ACuTe Heart Failure -Thrombolysis in Myocardial Infarction 68 (DAPA ACT HF-TIMI 68)
Brief Title: Dapagliflozin and Effect on Cardiovascular Events in Acute Heart Failure -Thrombolysis in Myocardial Infarction 68 (DAPA ACT HF-TIMI 68)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The TIMI Study Group (Other)
Collaborators: AstraZeneca (Industry); Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1690C00078
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Acute Heart Failure; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dapagliflozin (Experimental): Dapagliflozin 10 mg administered orally once daily for 2 months
  Interventions: Drug: Dapagliflozin
- Placebo (Placebo Comparator): Matching placebo administered orally once daily for 2 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — Dapagliflozin
  Arms: Dapagliflozin
Drug: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
This is an international, multicenter, parallel-group, randomized, double-blind, placebo-controlled trial in patients who have been stabilized during hospitalization for acute heart failure, evaluating the effect of in-hospital initiation of dapagliflozin versus placebo on the clinical outcome of cardiovascular death or worsening heart failure.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥18 years (male or female)
2. Currently hospitalized for AHF defined as meeting all the following criteria:

   1. Presentation with worsening symptoms of heart failure (e.g., worsening dyspnea or dyspnea at rest, progressive fatigue, rapid weight gain, worsening edema/abdominal distention/anasarca)
   2. Objective signs or diagnostic testing consistent with volume overload (e.g., jugular venous distension, pulmonary basilar crackles, S3 gallop, ascites, hepatomegaly, peripheral edema, radiological evidence of pulmonary congestion, noninvasive or invasive hemodynamic evidence of elevated filling pressures)
   3. Intensification of AHF therapy during admission defined as at least one of the following:

   i. Augmentation of oral diuretic therapy [e.g., ≥2x outpatient regimen dose, addition of a second diuretic agent, or new initiation of diuretic therapy in a previously naïve patient] ii. Initiation of intravenous diuretic therapy iii. Initiation of intravenous vasoactive agent (e.g., inotrope or vasodilator)
3. Left ventricular ejection fraction (LVEF) measured within the past 12 months (including during the current hospitalization)
4. Elevated NT-proBNP or BNP during current hospitalization:

   1. For patients with LVEF ≤40%: NT-proBNP ≥1600 pg/mL or BNP ≥400 pg/mL (NT-proBNP ≥2400 pg/mL or BNP ≥600 pg/mL if patient in atrial fibrillation or atrial flutter)
   2. For patients with LVEF >40%: NT-proBNP ≥1200 pg/mL or BNP ≥300 pg/mL (NT-proBNP ≥1800 pg/mL or BNP ≥450 pg/mL if patient in atrial fibrillation or atrial flutter)
5. Eligible patients will be randomized no earlier than 24 hours and up to 14 days after presentation while still hospitalized once they have been stabilized, as defined by:

   1. No increase (i.e., intensification) in the dose of intravenous diuretics during the 12 hours prior to randomization
   2. No use of intravenous vasodilators or inotropes during the 24 hours prior to randomization

Exclusion Criteria

1. Symptomatic hypotension in the past 24 hours
2. Concurrent use of two or more intravenous inotropic agents during the index hospitalization
3. eGFR <25 ml/min/1.73 m2 as measured by the CKD-EPI equation at screening or rapidly progressive renal disease
4. Current use of an SGLT2 inhibitor
5. Prior intolerance of SGLT2 inhibitors
6. Type 1 diabetes mellitus or history of diabetic ketoacidosis
7. (Only applies to patients with T2DM who are on insulin and/or a sulfonylurea) History of recurrent major hypoglycemia (i.e., resulting in severe impairment in consciousness or behavior, or requiring emergency external assistance)
8. Implantation of a cardiac resynchronization therapy (CRT) device or valve repair or replacement within 30 days prior to randomization or intent to do so during the trial
9. ST-segment elevation myocardial infarction or coronary revascularization (percutaneous coronary intervention or coronary artery bypass grafting) within 30 days prior to randomization or intent to undergo coronary revascularization during the trial
10. Untreated sustained ventricular arrhythmias or Mobitz type II or third-degree heart block (i.e., without an ICD or pacemaker, respectively)
11. History of heart transplantation or current transplant listing; mechanical circulatory support use (either durable or temporary) during the index hospitalization
12. History of heart failure due to restrictive or infiltrative cardiomyopathy, active myocarditis, constrictive pericarditis, hypertrophic (obstructive) cardiomyopathy, uncorrected primary valvular disease, complex congenital heart disease, or heart failure felt to be due to a transient process (e.g., stress [takotsubo] cardiomyopathy, tachycardia-induced cardiomyopathy) expected to resolve within 2 months.
13. History of end-stage liver disease
14. Women of child-bearing potential (unless using adequate contraception) or currently breastfeeding
15. Current participation in a clinical trial with an unlicensed drug or device
16. Study staff or their family members
17. Any condition that, in the opinion of the investigator, would make trial participation not in the best interest of the subject, or would compromise compliance with the trial protocol (e.g., active severe infection, active malignancy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2401 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Cardiovascular (CV) death or worsening heart failure | 2 months
  Time to first occurrence of CV death or worsening heart failure

SECONDARY OUTCOMES:
Composite CV death, rehospitalization for heart failure, urgent heart failure visit | 2 months
  Time to first occurrence of composite of CV death, rehospitalization for heart failure, or urgent heart failure visit
Composite CV death, rehospitalization for heart failure | 2 months
  Time to first occurrence of composite of CV death or rehospitalization for heart failure
Rehospitalization for heart failure, urgent heart failure visit | 2 months
  Time to first occurrence of rehospitalization for heart failure or urgent heart failure visit
Readmission | 2 months
  Readmission within 30 days of hospital discharge
CV death | 2 months
  Time to CV death
Death | 2 months
  Time to death

OTHER OUTCOMES:
Symptomatic hypotension | 2 months
  Symptomatic hypotension leading to hospitalization or study drug discontinuation
Worsening renal function | 2 months
  Worsening renal function resulting in at least a doubling of serum creatinine (sCr), hospitalization, study drug discontinuation, dialysis, or renal death

CONTACTS AND LOCATIONS:
Locations (1):
- TIMI Study Group, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berg DD, Patel SM, Haller PM, Cange AL, Palazzolo MG, Bellavia A, Kuder JF, Desai AS, Inzucchi SE, McMurray JJV, O'Meara E, Verma S, Belohlavek J, Drozdz J, Merkely B, Ogunniyi MO, Drasnar T, Izzo JL, Sarman B, McGinty JE, Ramanathan K, Mulkay AJ, Przybylski A, Ruff CT, O'Donoghue ML, Murphy SA, Sabatine MS, Wiviott SD; DAPA ACT HF-TIMI 68 Trial Committees and Investigators. Dapagliflozin in Patients Hospitalized for Heart Failure: Primary Results of the DAPA ACT HF-TIMI 68 Randomized Clinical Trial and Meta-Analysis of Sodium-Glucose Cotransporter-2 Inhibitors in Patients Hospitalized for Heart Failure. Circulation. 2025 Nov 18;152(20):1411-1422. doi: 10.1161/CIRCULATIONAHA.125.076575. Epub 2025 Aug 29. PMID 40884036
- [Derived] Berg DD, Patel SM, Haller PM, Belohlavek J, Desai AS, Drozdz J, Inzucchi SE, McMurray JJV, Merkely B, O'Meara E, Verma S, Cange AL, Murphy SA, Sabatine MS, Wiviott SD. Rationale and Design of the Dapagliflozin Effect on Cardiovascular Events in Acute Heart Failure (DAPA ACT HF)-TIMI 68 Trial. JACC Heart Fail. 2025 May;13(5):829-839. doi: 10.1016/j.jchf.2025.03.014. PMID 40335233